CLINICAL TRIAL: NCT04585802
Title: Expansion and Reevaluation of the Implicit Association Test in Suicide Ideators and Suicide Attempters
Acronym: IAT-S
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: University Hospital of Psychiatry, Department Neuropsychopharmacology and Brain Imaging (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-01410
Record Dates: First submitted 2020-09-23; First posted 2020-10-14 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Suicidal Ideation; Suicide Attempt
Keywords: Implicit Association Test
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Suicide Attempters (1): patients with a suicide attempt
- Suicide Ideators (2): patients with suicidal ideation
- Clinical Control Group (3): patients without suicide attempt and without suicide ideation
- Healthy Control Group (4): persons without suicide attempt and without suicide ideation, who do not have a psychiatric disorder

SUMMARY:
A new approach to investigate suicidal processes belongs to the broader neurocognitive picture and are so-called implicit associations. In dual process models of information processing a second functioning mode, the automatic processing mode, complements the conscious processing. Suicidal persons tend to have a stronger implicit association with "death" than non-suicidal persons. In this study, implicit associations between different unconscious cognitive constructs are compared among suicidal and non-suicidal patients. Therefore, an adapted version of the computer-based reaction time task (IAT-S) will be used.

Four different versions of IATs are tested in this study. In the first version the implicit association between "self / others" and "death / life" is assessed (1). The second and third version measures the emotional evaluation of "death" (2) and "life" (3). In addition, in the fourth version the implicit association between death / life and internal / external locus of control is assessed (4).

The implicit associations of these four IAT-S versions are compared between three groups: patients with suicidal behavior, patients with suicidal ideation, and a clinical group without previous suicide attempts and without suicidal ideation.

The following hypotheses are made: in all four versions of the IAT-S, patients with previous suicidal behavior will have stronger implicit associations: between "self" and "death" as well as "death" and "internal locus of control" compared to all other groups. With a more "positive" evaluation of "death" and a more "negative" evaluation of "life" than all other participants.

DETAILED DESCRIPTION:
In this study, four versions of the suicide-specific implicit association tests (IAT-S) are carried out. Previous studies have shown that suicidal persons have stronger associations between the constructs "self" and "death". Furthermore, the strength of these implicit associations increases the risk of suicidal behavior in the follow-up period of six months by a factor of six. In these previous studies, the implicit "self-death association" (the so-called death-identity bias) was investigated. This study will additionally examine an implicit emotional evaluation (death-evaluation-bias). Therefore, two new versions of the IAT-S, which measure how death vs. life are emotionally evaluated, are being tested. In addition, a fourth version of the IAT-S was added and aims to clarify the implicit association between death / life and internal / external locus of control. Previous studies have shown that an internal locus of control is a protective factor and an external locus of control a risk factor for suicide attempts. In the present study, these four IAT-S versions are carried out with different groups of patients: patients with a suicide attempt (1), patients with suicide ideation (2) and patients with neither a suicide attempt nor suicide ideation (3). This cross sectional design allows us to test for group differences in regard to unconscious implicit associations. Hypothesis are described separately for each version of the IAT-S.

Death association: patients in group 1 will have a higher implicit association between self and death than patients in group 2 and that patients in group 2 have a significantly higher implicit association between self and death than patients in group 3.

Death evaluation: patients in group 1 will have more "positive" evaluations of "death" than patients in group 2 and patients in group 2 have a more "positive" evaluations of death than patients in group 3.

Locus of control: patients in group 1 will have a stronger association between internal locus of control and death (a) and external locus of control and life (b) than patients in group 2, and that patients in group 2 have a significantly stronger association between internal locus of control and death (a) and external locus of control and life (b) than patients in group 3.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Ability and willingness to participate in the study
* Ability to give consent

Exclusion Criteria:

* Foreign language
* Diagnostic criteria: Psychoses, strong cognitive impairments (e.g. dementia)

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients from the University Hospital of Psychiatry
Sampling Method: Probability Sample
Enrollment: 447 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Implicit Association Test (IAT) | One assessment at baseline after study information and informed consent was given
  The German version of the Suicide Implicit Association Test (Rath et al., 2018) is administered using a computer paradigm and is designed to measure implicit associations with death using D-values. D is an individual effect size assessment that reflects the comparative difficulty of performing the two response conditions of the IAT, with a value of 0 indicating that the tasks had equivalent performance (Greenwald et al., 2003). D has a theoretical minimum of -2 and maximum of +2 when blocks of the same size are compared (Nosek & Sriram, 2007). The more positive the D-values, the stronger the association between the "self" and "death" than between the "self" and "life".

SECONDARY OUTCOMES:
Suicide Behaviors Questionnaire - Revised | One assessment at baseline after study information and informed consent was given
  The Suicide Behaviors Questionnaire measures suicidal behavior in the past and consists of four items. Item scores range from 3 to 18 with higher scores indicating more suicidal behavior (Osman et al., 2001).
Beck Scale for Suicide Ideation (BSS) | One assessment at baseline after study information and informed consent was given
  The Beck-Scale for Suicide Ideation measures suicidal thinking and consists of 21 items. Item scores range from 0 to 42 with higher scores indicating more suicidal ideation (Beck & Steer, 1993; Kliem & Brähler, 2016).
Beck Depression Inventory (BDI-II) | One assessment at baseline after study information and informed consent was given
  The Beck Depression Inventory measures the severity of depression and consists of 21 items. Item scores range from 0 to 63 with higher scores indicating a higher intensity of depression (Beck, Steer & Brown, 1996).
Mee-Bunney Psychological Pain Assessment Scale (MBPPAS) | One assessment at baseline after study information and informed consent was given
  The Mee-Bunney Psychological Pain Assessment Scale measures psychological pain and consists of 10 items. Item scores range from 10 to 50 with higher scores indicating more psychological pain (Mee et al., 2011).
Positive Mental Health Scale (PMH-scale) | One assessment at baseline after study information and informed consent was given
  Positive Mental Health Scale measures positive mental health ans consists of 9 items. Item scores range from 9 to 36 with higher scores indicating more positive mental health (Lukat, Margraf, Lutz, van der Veld & Becker, 2016).
Internal External Locus of Control-4 (IE-4) | One assessment at baseline after study information and informed consent was given
  The IE-4 is a Scale for the Assessment of Locus of Control and consists of two subscales with two items each. For each subscale, the mean value of the two items is calculated, which can range from 1 to 5 with higher scores indication more internal/external locus of control (Kemper, Beierlein, Kovaleva, & Rammstedt, 2012).
Mini-International Neuropsychiatric Interview (M.I.N.I.) | One assessment at baseline after study information and informed consent was given
  The Mini-International Neuropsychiatric Interview is a brief structured diagnostic interview to assess the most common psychiatric disorders (Sheehan et al., 1998).

CONTACTS AND LOCATIONS:
Overall Officials: Anja C. Gysin-Maillart, PD, Principal Investigator — University of Bern
Locations (1):
- University Hospital of Psychiatry and Psychotherapy, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nock MK, Park JM, Finn CT, Deliberto TL, Dour HJ, Banaji MR. Measuring the suicidal mind: implicit cognition predicts suicidal behavior. Psychol Sci. 2010 Apr;21(4):511-7. doi: 10.1177/0956797610364762. Epub 2010 Mar 9. PMID 20424092
- [Background] Pearce CM, Martin G. Locus of control as an indicator of risk for suicidal behaviour among adolescents. Acta Psychiatr Scand. 1993 Dec;88(6):409-14. doi: 10.1111/j.1600-0447.1993.tb03482.x. PMID 8310847
- [Background] Rath D, Hallensleben N, Glaesmer H, Spangenberg L, Strauss M, Kersting A, Teismann T, Forkmann T. [Implicit Associations with Death: First Validation of the German Version of the Suicide Implicit Association Test (Suicide IAT)]. Psychother Psychosom Med Psychol. 2018 Mar;68(3-4):109-117. doi: 10.1055/s-0043-105070. Epub 2017 Jun 29. German. PMID 28718868
- [Background] Everall, RD, Altrows, KJ, Paulson, BL. Creating a Future: A Study of Resilience in Suicidal Female Adolescents. Journal of Counseling & Development. 2006; 84(4): 461-470.
- [Background] Osman A, Bagge CL, Gutierrez PM, Konick LC, Kopper BA, Barrios FX. The Suicidal Behaviors Questionnaire-Revised (SBQ-R): validation with clinical and nonclinical samples. Assessment. 2001 Dec;8(4):443-54. doi: 10.1177/107319110100800409. PMID 11785588
- [Background] Beck AT, Steer RA, Ball R, Ranieri W. Comparison of Beck Depression Inventories -IA and -II in psychiatric outpatients. J Pers Assess. 1996 Dec;67(3):588-97. doi: 10.1207/s15327752jpa6703_13. PMID 8991972
- [Background] Beck AT, Steer RA. BSI, Beck Scale for Suicide Ideation. Psychological Corporation. 1993.
- [Background] Kliem S, Brähler E. Beck-Hoffnungslosigkeits-Skala. Deutsche Fassung. Göttingen:Hogrefe. 2016.
- [Background] Mee S, Bunney BG, Bunney WE, Hetrick W, Potkin SG, Reist C. Assessment of psychological pain in major depressive episodes. J Psychiatr Res. 2011 Nov;45(11):1504-10. doi: 10.1016/j.jpsychires.2011.06.011. Epub 2011 Aug 9. PMID 21831397
- [Background] Lukat J, Margraf J, Lutz R, van der Veld WM, Becker ES. Psychometric properties of the Positive Mental Health Scale (PMH-scale). BMC Psychol. 2016 Feb 10;4:8. doi: 10.1186/s40359-016-0111-x. PMID 26865173
- [Background] Kemper CJ, Beierlein C, Kovaleva A, Rammstedt B. Eine Kurzskala zur Messung von Kontrollüberzeugung: Die Skala lnternale-Externale Kontrollüberzeugung-4 (IE-4). GESIS Working Papers.2012; 2(19).
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Nosek BA, Sriram N. Faulty assumptions: A comment on Blanton, Jaccard, Gonzales, and Christie (2006). J Exp Soc Psychol. 2007 May;43(3):393-398. doi: 10.1016/j.jesp.2006.10.018. PMID 18438456
- [Background] Greenwald AG, Nosek BA, Banaji MR. Understanding and using the implicit association test: I. An improved scoring algorithm. J Pers Soc Psychol. 2003 Aug;85(2):197-216. doi: 10.1037/0022-3514.85.2.197. PMID 12916565